CLINICAL TRIAL: NCT03039179
Title: Effectiveness of Polyurethane Foam in Preventing the Onset of Pressure Sores in a Pediatric Orthopedic Population: Randomized Controlled Trial
Brief Title: Polyurethane Foam on the Heel for Prevention in Children
Acronym: SCHIUMABIMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0024520
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2017-04

CONDITIONS: Flat Foot; Pressure Ulcer
MeSH Terms: conditions — Flatfoot; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyurethane foam (Experimental)
  Interventions: Device: polyurethane foam dress
- standard care (No Intervention): Only application of the Walker in the immediate postoperative period.

INTERVENTIONS:
Device: polyurethane foam dress — Application of the polyurethane foam dress at the heel in the immediate postoperative period before applied the Walker
  Arms: Polyurethane foam

SUMMARY:
The post-operative treatment of pediatric patients operated for the correction of flat foot, sees today the use of preformed leg-foot splint (Walker) as an alternative to the application of plaster casts. The change of the immobilization system has led to the appearance of problems of tolerability in particular in the skin. The aim of the study is to assess whether by placing a polyurethane foam dress at the heel in the immediate postoperative period until removal of the Walker, the rate of skin lesion and pain is reduced.

ELIGIBILITY:
Inclusion Criteria:

* Children aged > 3 years underwent surgery for flat foot
* Children with intact skin at the heel

Exclusion Criteria:

* Caregivers who cannot speak Italian
* Those who refuse to give their consent to take part in the study
* Patients with lower limb casts after surgery

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Guerra, RN, Principal Investigator — Istituto Ortopedico Rizzoli

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began on May 2014 and ended in May 2015 when the eighties patient was enrolled.
Period: Overall Study
Arm/Group | Polyurethane Foam | Standard Care
Started | 38 | 42
Completed | 38 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polyurethane Foam | Standard Care | Total
Number analyzed (Participants) | 38 | 42 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.79 (1.27) | 11.64 (1.44) | 11.71 (1.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 23 | 26 | 49
type of surgery:Calcaneal Osteotomy [Count of Participants; unit: Participants] | 37 | 39 | 76
type of analgesia:peripheral nerve blocks analgesia [Count of Participants; unit: Participants] | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Heel Pressure Sores (Numbers of Participants With Heel Pressure Sores)
Description: Numbers of Participants With Heel Pressure Sores of all grade Detected According to the Classification of the Scale of the National Pressure Ulcer Advisory Panel -N.P.U.A.P.: Grade 1: Non-blanchable erythema of intact skin. Discoloration of the skin, warmth, oedema, induration or hardness may also be used as indicators, particularly in individuals with darker skin. Grade 2: Partial thickness skin loss involving epidermis, dermis, or both. The ulcer is superficial and presents clinically as an abrasion or blister. Grade 3: Full thickness skin loss involving damage to or necrosis of subcutaneous tissue that may extend down to, but not through, underlying fascia. Grade 4: Extensive destruction, tissue necrosis, or damage to muscle, bone, or supporting structures with or without full thickness skin loss.
Time Frame: every day until discharge (expected average of 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Polyurethane Foam | Standard Care
Number analyzed (Participants) | 38 | 42
Participants | 17 | 21

2. Secondary Outcome: Pain (Score on the "Numeric Rating Scale")
Description: Pain Score on the "Numeric Rating Scale" > 3. The scale had values from 0 to 10 where zero represented no pain and 10 the worst possible pain. More than 3 means pain.
Time Frame: up to the first 3 days post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Polyurethane Foam | Standard Care
Number analyzed (Participants) | 38 | 42
Participants | 26 | 25

ADVERSE EVENTS:
Arm/Group | Polyurethane Foam | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/42
Other Adverse Events (participants affected / at risk) | 0/38 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No